CLINICAL TRIAL: NCT01465815
Title: Phase I/II Study of Postoperative Adjuvant Chemoradiation for cSCCHN
Brief Title: Phase I/II Study of Postoperative Adjuvant Chemoradiation for Advanced-Stage Cutaneous Squamous Cell Carcinoma of the Head and Neck (cSCCHN)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug manufacturer, Astellas Pharma, informed us that safety and efficacy of Erlotinib and OSI-906 in other oncology studies was determined to be unfavorable.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6901 (5466); NCI-2011-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-26; First posted 2011-11-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Recurrent Skin Cancer; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Squamous Cell Carcinoma of the Skin; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity
MeSH Terms: conditions — Skin Neoplasms | interventions — Erlotinib Hydrochloride; 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment (adjuvant enzyme inhibitor and radiation therapy) (Experimental): Optional non-therapeutic (biomarker) portion: Patients are randomized to 1 of 3 treatment arms.
  Arm A: Patients receive erlotinib hydrochloride PO QD and linsitinib PO BID on days 1-7 or 1-14.
  Treatment continues until 1 day before planned surgical resection (for up to 28 days if surgery is delayed).
  Therapeutic portion: This is a phase I dose-escalation study of linsitinib followed by a phase II study.
  Patients undergo standard QD conventional radiotherapy at the discretion of the treating physician. Patients receive concurrent linsitinib PO BID and erlotinib hydrochloride PO QD during the entire course of radiation in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: linsitinib; Radiation: radiation therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Erlotinib and Placebo (Sugar Pill) (Experimental): Arm B: Patients receive erlotinib hydrochloride PO QD and placebo PO QD or BID on days 1-7 or 1-14.
  Treatment continues until 1 day before planned surgical resection (for up to 28 days if surgery is delayed).
  Therapeutic portion: This is a phase I dose-escalation study of linsitinib followed by a phase II study.
  Patients undergo standard QD conventional radiotherapy at the discretion of the treating physician. Patients receive concurrent linsitinib PO BID and erlotinib hydrochloride PO QD during the entire course of radiation in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: placebo
- OSI-906 and Placebo (Sugar Pill) (Experimental): Arm C: Patients receive linsitinib PO BID and placebo PO QD or BID on days 1-7 or 1-14.
  Treatment continues until 1 day before planned surgical resection (for up to 28 days if surgery is delayed).
  Therapeutic portion: This is a phase I dose-escalation study of linsitinib followed by a phase II study.
  Patients undergo standard QD conventional radiotherapy at the discretion of the treating physician. Patients receive concurrent linsitinib PO BID and erlotinib hydrochloride PO QD during the entire course of radiation in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: linsitinib; Drug: placebo

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
  Arms: Erlotinib and Placebo (Sugar Pill); Treatment (adjuvant enzyme inhibitor and radiation therapy)
Drug: linsitinib — Given PO
  Other Names: OSI-906
  Arms: OSI-906 and Placebo (Sugar Pill); Treatment (adjuvant enzyme inhibitor and radiation therapy)
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Erlotinib and Placebo (Sugar Pill); OSI-906 and Placebo (Sugar Pill)
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
  Arms: Treatment (adjuvant enzyme inhibitor and radiation therapy)
Procedure: therapeutic conventional surgery — Undergo planned surgery
  Arms: Treatment (adjuvant enzyme inhibitor and radiation therapy)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Treatment (adjuvant enzyme inhibitor and radiation therapy)

SUMMARY:
This phase I/II trial studies the side effects and best dose of linsitinib when given together with erlotinib hydrochloride and radiation therapy after surgery in treating patients with advanced or recurrent head and neck cancer. Erlotinib hydrochloride and linsitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy together with erlotinib hydrochloride and linsitinib may kill more tumor cells. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the MTD (maximally tolerated dose) of OSI-906 (linsitinib) when used in combination with erlotinib (erlotinib hydrochloride) and radiation therapy after surgery for advanced-stage cutaneous squamous cell carcinoma of the head and neck (cSCCHN). (Phase I) II. To estimate the 2-year overall survival (OS) compared to historical controls. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of OSI-906 in combination with erlotinib and radiation therapy after surgery for advanced-stage cSCCHN.

II. To estimate the 2-year disease specific and disease free survival. III. To determine the time to recurrence and patterns of failure. IV. To evaluate the effects of short-term preoperative treatment with erlotinib and OSI-906 on the expression epidermal growth factor receptor (EGFR), insulin-like growth factor 1 receptor (IGF-1R) and parallel or downstream molecular targets in cSCCHN in one third of the patients.

OUTLINE:

Optional non-therapeutic (biomarker) portion: Patients are randomized to 1 of 3 treatment arms.

Arm A: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) and linsitinib PO twice daily (BID) on days 1-7 or 1-14.

Arm B: Patients receive erlotinib hydrochloride PO QD and placebo PO QD or BID on days 1-7 or 1-14.

Arm C: Patients receive linsitinib PO BID and placebo PO QD or BID on days 1-7 or 1-14.

Treatment continues until 1 day before planned surgical resection (for up to 28 days if surgery is delayed).

Therapeutic portion: This is a phase I dose-escalation study of linsitinib followed by a phase II study.

Patients undergo standard QD conventional radiotherapy at the discretion of the treating physician. Patients receive concurrent linsitinib PO BID and erlotinib hydrochloride PO QD during the entire course of radiation in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 and 12 weeks, every 12-16 weeks for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have primary or recurrent advanced-stage (III/IV) squamous cell carcinoma of the skin of the face, ear, scalp or neck or of the lip
* A biopsy or preserved representative tumor block is required to confirm the diagnosis
* Patients must be surgical candidates with resectable disease; macroscopic complete resection of all tumor must be planned with curative intent
* Patients must be willing to receive postoperative radiation therapy and treatment with study drugs
* Both men and women and members of all races and ethnic groups will be included
* Life expectancy of greater than 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/microliter(uL)
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/uL
* International normalized ratio (INR) < institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x institutional ULN
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 2.5 X institutional ULN
* Creatinine =< 1.5 X institutional ULN
* Fasting blood glucose < 125 mg/dL at baseline
* Patients-both males and females-with reproductive potential (i.e., menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study; women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known distant metastasis
* Patients who have had prior radiation treatment of the index cancer or area of disease
* Patients who have received any other investigational medication within 6 weeks of enrollment, or who are scheduled to receive an investigational drug during the course of the study
* Prior treatment with EGFR inhibitor for index cancer
* Prior treatment with an IGF-1R antagonist (small molecule inhibitor or antibody)
* Breast-feeding, pregnancy or of childbearing potential (including less than two years postmenopausal) and unable to confirm adequate contraception due to possible risk to fetus or infant
* Insulin-dependent and non-insulin dependent diabetes mellitus including any metformin or insulin use on an ongoing basis prior to enrollment
* Known severe hypersensitivity to erlotinib, other small molecule inhibitors of EGFR, or its excipients
* Hepatitis B or C infection (acute or chronic), known human immunodeficiency virus (HIV), or active uncontrolled infection, because of possible risk of lethal infection when treated with marrow suppressive therapy
* History of uncontrolled cardiac disease such as unstable angina pectoris, myocardial infarction within prior 6 months, untreated coronary artery disease, uncontrolled congestive heart failure, or cardiomyopathy with decreased ejection fraction
* Uncontrolled peptic or gastric ulcer disease or gastrointestinal bleeding within prior 6 months
* Corrected QT interval (QTc) > 450 msec; congenital long QT syndrome or previous history of QTc prolongation as a result from other medication
* Presence of left bundle branch block (LBBB); QTc with Bazett's correction that is unmeasurable, or >= 450 msec on screening electrocardiogram (EKG)
* Any concomitant medication that may cause QTc prolongation or concomitant medication that is associated with Torsades de Pointes
* Psychiatric illness/social situations that would limit compliance with study requirements
* Active smokers unwilling to quit smoking during treatment
* Use of the potent cytochrome P450 3A4 (CYP3A4) and cytochrome P450 1A2 (CYP1A2) inhibitors is not allowed; other less potent CYP3A4 and CYP1A2 inhibitors/inducers are not excluded
* Participation in another investigational trial while on this study is not allowed
* History of poorly controlled gastrointestinal disorders including acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, Crohn's disease, ulcerative colitis or other diseases which have the potential for bowel perforation
* Other malignancies except for resected cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with overall survival(OS) after two years of treatment (Phase II) | Up to 2 years
  The 2-year OS and 95% confidence interval will be determined using Kaplan-Meier method.
The maximum tolerated dose (MTD) of linsitinib when used in combination with erlotinib hydrochloride and radiation therapy (phase 1) | up to 24 months
  The MTD of linsitinib when used in combination with erlotinib hydrochloride and radiation therapy will be determined using a standard 3x3 dose-escalation scheme. The dose limiting toxicity (DLT) will be defined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.02). DLT is defined as any grade 3 non-hematologic toxicity attributed to treatment or grade 4 hematologic toxicity, neutropenic fever requiring hospitalization, or treatment delay due to hematologic toxicity.
The maximum tolerated dose (MTD) of linsitinib when used in combination with erlotinib hydrochloride and radiation therapy (phase 1) | Up to 5 years
  The MTD of linsitinib when used in combination with erlotinib hydrochloride and radiation therapy will be determined using a standard 3x3 dose-escalation scheme. The dose limiting toxicity (DLT) will be defined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events CTCAE (v4.02). DLT is defined as any grade 3 non-hematologic toxicity attributed to treatment or grade 4 hematologic toxicity, neutropenic fever requiring hospitalization, or treatment delay due to hematologic toxicity.

SECONDARY OUTCOMES:
Number of participants with disease free survival | At 2 years
Time to recurrence and patterns of failure | Up to 2 years
Effects of short-term preoperative treatment with erlotinib hydrochloride and linsitinib on the expression EGFR, IGF-1R and parallel or downstream molecular targets in cSCCHN in one third of the patients | From baseline to time of surgery (after 7-14 days of study drug administration)
Number of adverse events observed from linsitinib in combination with erlotinib hydrochloride and radiation therapy. | After completion of study therapy at 6 and 12 weeks
Number of adverse events observed from linsitinib in combination with erlotinib hydrochloride and radiation therapy | Every 12-16 weeks for 2 years
Number of adverse events observed from linsitinib in combination with erlotinib hydrochloride and radiation therapy | Every 6 months for 3 years and then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Neil Gross, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States